CLINICAL TRIAL: NCT05875051
Title: Effects of Reduced-exertion High-intensity Training Versus Short Moderate Intensity Training on Functional Capacity and Physical Activity Enjoyment in Sedentary Young Women A Randomized Trial
Brief Title: REHIT Versus SMIT in Sedentary Young Women
Acronym: REHIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Elena Marques-Sule, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 035/3/20
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Sedentary Behavior
Keywords: High-intensity training; Moderate intensity training; Sedentary young women
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to treatment group allocation. The blinded assessor will collect all baseline and post-intervention measures and enter data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced-exertion high intensity training group (Experimental): The REHIT part will consist of maximum cycling sprints of all-out exercise at 100% of the HRmax, increasing for up to 10 seconds, 15 seconds on week two and 20 seconds on week three.
  Interventions: Other: Reduced-exertion high intensity training
- Short moderate intensity training group (Active Comparator): The SMIT part of the session will consist of 6 minutes of moderate intensity exercise at 60-70% HRmax.
  Interventions: Other: Short moderate intensity training

INTERVENTIONS:
Other: Reduced-exertion high intensity training — The intervention of the REHIT group will consist of three parts: i) 3 minutes of warm-up part at 50% of HRmax obtained in the effort test; ii) 3 min 20 sec to 3 min 40 sec of REHIT; and iii) 3 minutes of cool-down at 50% of HRmax obtained in the effort test. The REHIT part will consist of maximum cycling sprints of all-out exercise at 100% of the HRmax, increasing for up to 10 seconds, 15 seconds on week two and 20 seconds on week three. Then, 3 minutes of active rest at 50% of HRmax. Finally, 10 seconds of all-out exercise at 100% of the HRmax, rising to 15 seconds on week two and 20 seconds on week three.
  Arms: Reduced-exertion high intensity training group
Other: Short moderate intensity training — The SMIT group will receive a short moderate-intensity training with the same warm-up and cool-down exercises as the REHIT group. In addition, the main part of the session consisted of 6 minutes of moderate intensity exercise at 60-70% HRmax obtained in the effort test. In addition, the main part of the session increases 3 min every week as 6 min for the first 2 weeks, 9 min for the 3rd and 4th weeks, and 12 min for the last two weeks.
  Arms: Short moderate intensity training group

SUMMARY:
Reduced-exertion high-intensity training (REHIT) is a novel form of exercise known for being non-classical, time-efficient, and effective on different populations. However, REHIT was scarcely tested on sedentary women with mortality risks. The aim of the study is to compare the effects of REHIT versus short moderate-intensity training (SMIT) on functional capacity, resting heart rate (RHR), and activity enjoyment in sedentary young women.

DETAILED DESCRIPTION:
The aim of the study is to compare the effects of reduced-exertion high-intensity training (REHIT) versus short moderate-intensity training (SMIT) on functional capacity, resting heart rate (RHR), and activity enjoyment in sedentary young women. Therefore, sedentary young women will be randomly allocated to either a: i) REHIT group or ii) SMIT group. Both groups will perform an intervention over 6 weeks duration for 10 minutes each session for 2 sessions/week, but with different intensities (REHIT or SMIT). Both forms of exercise will be conducted on a cycle ergometer with the subjects monitored throughout the intervention. Before and after the 3-week intervention, functional capacity (6-minute walking test) and RHR will be measured. Additionally, physical activity enjoyment (Physical Activity Enjoyment Scale) will be assessed after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women.
* Age between 18 and 25 years old.
* Those who score a low physical activity level (< 600 METS min/week) in the International Physical Activity Questionnaire-short form.

Exclusion Criteria:

* Women who suffer from musculoskeletal.
* Women who suffer from neurological diseases.
* Those who are taking medications.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Functional capacity | Baseline
  It will be measured using the 6-minutes walking test (6MWT). Participants will be instructed to walk as quickly as possible along a 30-meter hallway for a duration of six minutes without running. Then, the distance in meters they cover will be registered. The greater the number of meters run, the better the functional capacity.
Functional capacity | After the intervention (3 weeks)
  It will be measured using the 6-minutes walking test (6MWT). Participants will be instructed to walk as quickly as possible along a 30-meter hallway for a duration of six minutes without running. Then, the distance in meters they cover will be registered. The greater the number of meters run, the better the functional capacity.

SECONDARY OUTCOMES:
Resting heart rate | Baseline
  It will be measured with a patient monitor (ProAct PC-3000 Patient Monitor, Medisave, UK).
Resting heart rate | After the intervention (3 weeks)
  It will be measured with a patient monitor (ProAct PC-3000 Patient Monitor, Medisave, UK).
Physical activity enjoyment | Baseline
  To assess enjoyment, a modified version of the Physical Activity Enjoyment Scale (PACES) will be used. In this questionnaire, 17 items are scored on a 7-point bipolar scale, with an overall enjoyment score ranging from 17 (not enjoyable) to 68 (neutral) and 119 (enjoyable).
Physical activity enjoyment | After the intervention (3 weeks)
  To assess enjoyment, a modified version of the Physical Activity Enjoyment Scale (PACES) will be used. In this questionnaire, 17 items are scored on a 7-point bipolar scale, with an overall enjoyment score ranging from 17 (not enjoyable) to 68 (neutral) and 119 (enjoyable).

CONTACTS AND LOCATIONS:
Overall Officials: Elena Marqués Sulé, PhD, Principal Investigator — Univeristy of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Metcalfe RS, Atef H, Mackintosh K, McNarry M, Ryde G, Hill DM, Vollaard NBJ. Time-efficient and computer-guided sprint interval exercise training for improving health in the workplace: a randomised mixed-methods feasibility study in office-based employees. BMC Public Health. 2020 Mar 12;20(1):313. doi: 10.1186/s12889-020-8444-z. PMID 32164631
- [Background] Ramirez-Velez R, Hernandez-Quinones PA, Tordecilla-Sanders A, Alvarez C, Ramirez-Campillo R, Izquierdo M, Correa-Bautista JE, Garcia-Hermoso A, Garcia RG. Effectiveness of HIIT compared to moderate continuous training in improving vascular parameters in inactive adults. Lipids Health Dis. 2019 Feb 4;18(1):42. doi: 10.1186/s12944-019-0981-z. PMID 30717757
- [Background] Metcalfe RS, Tardif N, Thompson D, Vollaard NB. Changes in aerobic capacity and glycaemic control in response to reduced-exertion high-intensity interval training (REHIT) are not different between sedentary men and women. Appl Physiol Nutr Metab. 2016 Nov;41(11):1117-1123. doi: 10.1139/apnm-2016-0253. Epub 2016 Jul 7. PMID 27753506
- [Derived] Bahey El-Deen HA, Atef H, Munoz-Gomez E, Moreno-Segura N, ElZalabany S, Alanazi R, Alruwili W, Alruwili S, Sultan S, Marques-Sule E. Effects of reduced-exertion high-intensity training versus short moderate-intensity continuous training on biomarkers of mortality risk in sedentary women: A randomized clinical trial. J Bodyw Mov Ther. 2025 Jun;42:710-714. doi: 10.1016/j.jbmt.2025.01.056. Epub 2025 Feb 2. PMID 40325745